CLINICAL TRIAL: NCT05305651
Title: Prospective Cohort Study to Monitor the Emergence of SARS-CoV-2 Spike Viral Variants in Immunocompromised Non-hospitalized Patients Exposed to Sotrovimab in Great Britain: LUNAR Study
Brief Title: Study to Monitor the Occurrence of Viral Variants in Patients With Compromised Immune Systems Being Treated for COVID-19
Acronym: LUNAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 218407
Record Dates: First submitted 2022-03-30; First posted 2022-03-31 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: COVID-19
Keywords: SARS CoV-2; LUNAR; Coronavirus disease 2019 (COVID-19); Pandemic; Sotrovimab; Monoclonal antibody; Immunocompromised (IC)
MeSH Terms: conditions — COVID-19 | interventions — sotrovimab

STUDY DESIGN:
Intervention Model Description: This study is a prospective cohort study which will enroll IC non-hospitalized participants receiving sotrovimab treatment as per standard of clinical care for COVID-19 in sentinel sites.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants receiving Sotrovimab (Experimental): Immunocompromised non-hospitalized participants will receive sotrovimab as standard of clinical care for COVID-19 in sentinel sites
  Interventions: Drug: Sotrovimab

INTERVENTIONS:
Drug: Sotrovimab — Sotrovimab dose and administration per standard of clinical care

SUMMARY:
Sotrovimab binds to a conserved epitope on the severe acute respiratory syndrome coronavirus (SARS-CoV) and SARS-CoV-2 spike protein outside the receptor-binding motif and has been shown to reduce the risk of hospitalization and/or death when administered as early treatment in non-hospitalized patients that are at risk for progression to severe disease. Immunocompromised (IC) patients are prioritized to receive early treatment for COVID-19 as they are at high risk of disease progression, and because of their potential for prolonged viral shedding and the resulting increased risk of emergent viral mutations and potential onward community transmission.

This genomic surveillance study will aim to describe changes in the SARS-CoV-2 spike protein observed in IC participants receiving sotrovimab as standard of clinical care in sentinel sites at a national level to assess potential emergence of viral variants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be adult and of greater than or equal to (>=) 18 years of age or older at the time of consent
* Participants must be immunocompromised (IC) population eligible to receive sotrovimab
* A positive polymerase chain reaction (PCR) or antigen test for SARS-CoV-2 through clinical testing or routine screening undertaken as part of clinical management
* Prescribed treatment with sotrovimab as standard of clinical care
* Able to provide informed consent and willing to adhere to study-related procedures

Exclusion Criteria:

* Participants who require hospitalization (related or not to COVID-19) at baseline
* Participants who initiated sotrovimab therapy in inpatient settings
* Participants unable to perform nasal/oropharyngeal sample collection
* Blinded participants from other COVID-19 related trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United Kingdom (7):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, EdgbastonBirmingham
  - GSK Investigational Site, London
  - GSK Investigational Site, Middlesbrough
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Case JB, Mackin S, Errico JM, Chong Z, Madden EA, Whitener B, Guarino B, Schmid MA, Rosenthal K, Ren K, Dang HV, Snell G, Jung A, Droit L, Handley SA, Halfmann PJ, Kawaoka Y, Crowe JE Jr, Fremont DH, Virgin HW, Loo YM, Esser MT, Purcell LA, Corti D, Diamond MS. Resilience of S309 and AZD7442 monoclonal antibody treatments against infection by SARS-CoV-2 Omicron lineage strains. Nat Commun. 2022 Jul 2;13(1):3824. doi: 10.1038/s41467-022-31615-7. PMID 35780162

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective cohort study amongst immunocompromised non-hospitalized participants treated with sotrovimab as part of standard clinical care to monitor the emergence of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) spike viral variants.
Pre-assignment Details: A total of 217 participants were enrolled in this study.
Groups:
- Sotrovimab 500 mg IV: Immunocompromised non-hospitalized participants were treated with sotrovimab 500 milligram (mg) intravenously (IV) as a standard of clinical care for Coronavirus Disease 2019 (COVID-19).
Period: Overall Study
Arm/Group | Sotrovimab 500 mg IV
Started | 217
Completed | 208
Not Completed | 9
Not completed — Death | 1
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Sotrovimab 500 mg IV
Number analyzed (Participants) | 217
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.5 (15.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123
  Male | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Few race categories (with 0<n<11) are combined into one 'De-identified' category to maintain participant confidentiality and privacy, as they could lead to participant re-identification.
  Participants
    White | 49
    White - White/Caucasian/European Heritage | 139
    De-identified | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Amino Acid Substitutions Greater Than (>) 5 Percent (%) and >50% Allelic Frequency in the Sotrovimab Epitope at Day 7
Description: SARS-CoV-2 spike analysis was carried out by nucleotide sequencing of the SARS-CoV-2 spike protein by Next generation sequencing (NGS) analysis of participant nasal/oropharyngeal swab samples. The nucleotide sequences were translated, and the amino acid (AA) sequences aligned and compared to a reference sequence. Treatment emergent (TE) substitutions are defined as AA differences in a post-Baseline sample that were not present at Baseline at the defined threshold for minority and consensus analysis. The epitope is part of the spike protein, and it was analyzed separately from the rest of spike. The number of participants with TE substitutions in the sotrovimab epitope reflects participants that had a TE change in the spike protein at the sotrovimab epitope position only. AA substitutions compared to the reference strain are presented at Day 7.
Time Frame: At Day 7
Population: The Safety Set included all participants who were enrolled and exposed to study intervention. Only those participants with Paired Sequences were included in the analysis. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab 500 mg IV
Number analyzed (Participants) | 153
Participants
  AA substitutions >5% allelic frequency | 38
  AA substitutions >50% allelic frequency | 12

2. Primary Outcome: Number of Participants With Treatment Emergent Amino Acid Substitutions >5% and >50% Allelic Frequency in the Sotrovimab Epitope at Day 14
Description: SARS-CoV-2 spike analysis was carried out by nucleotide sequencing of the SARS-CoV-2 spike protein by NGS analysis of participant nasal/oropharyngeal swab samples. The nucleotide sequences were translated, and AA sequences aligned and compared to a reference sequence. Treatment emergent (TE) substitutions are defined as AA differences in a post-Baseline sample that were not present at Baseline at the defined threshold for minority and consensus analysis. The epitope is part of the spike protein, and it was analyzed separately from the rest of spike. The number of participants with TE substitutions in the sotrovimab epitope reflects participants that had a TE change in the spike protein at the sotrovimab epitope position only. AA substitutions compared to the reference strain are presented at Day 14.
Time Frame: At Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab 500 mg IV
Number analyzed (Participants) | 71
Participants
  AA substitutions >5% allelic frequency | 18
  AA substitutions >50% allelic frequency | 11

3. Primary Outcome: Number of Participants With Treatment Emergent Amino Acid Substitutions >5% and >50% Allelic Frequency in the Sotrovimab Epitope at Day 28
Description: SARS-CoV-2 spike analysis was carried out by nucleotide sequencing of the SARS-CoV-2 spike protein by NGS analysis of participant nasal/oropharyngeal swab samples. The nucleotide sequences were translated, and AA sequences aligned and compared to a reference sequence. Treatment emergent (TE) substitutions are defined as AA differences in a post-Baseline sample that were not present at Baseline at the defined threshold for minority and consensus analysis. The epitope is part of the spike protein, and it was analyzed separately from the rest of spike. The number of participants with TE substitutions in the sotrovimab epitope reflects participants that had a TE change in the spike protein at the sotrovimab epitope position only. AA substitutions compared to the reference strain are presented at Day 28.
Time Frame: At Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab 500 mg IV
Number analyzed (Participants) | 33
Participants
  AA substitutions >5% allelic frequency | 11
  AA substitutions >50% allelic frequency | 11

4. Primary Outcome: Number of Participants With Treatment Emergent Amino Acid Substitutions >5% and >50% Allelic Frequency in the Spike Protein at Day 7
Description: SARS-CoV-2 spike analysis was carried out by nucleotide sequencing of the SARS-CoV-2 spike protein by NGS analysis of participant nasal/oropharyngeal swab samples. The nucleotide sequences were translated, and the AA sequences aligned and compared to a reference sequence. Treatment emergent (TE) substitutions are defined as AA differences in a post-Baseline sample that were not present at Baseline at the defined threshold for minority and consensus analysis. The number of participants with TE substitutions in the spike protein reflects participants that had a TE change in the spike protein at any position including the sotrovimab epitope. AA substitutions compared to the reference strain are presented at Day 7.
Time Frame: At Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab 500 mg IV
Number analyzed (Participants) | 153
Participants
  AA substitutions >5% allelic frequency | 88
  AA substitutions >50% allelic frequency | 19

5. Primary Outcome: Number of Participants With Treatment Emergent Amino Acid Substitutions >5% and >50% Allelic Frequency in the Spike Protein at Day 14
Description: SARS-CoV-2 spike analysis was carried out by nucleotide sequencing of the SARS-CoV-2 spike protein by NGS analysis of participant nasal/oropharyngeal swab samples. The nucleotide sequences were translated, and the AA sequences aligned and compared to a reference sequence. Treatment emergent (TE) substitutions are defined as AA differences in a post-Baseline sample that were not present at Baseline at the defined threshold for minority and consensus analysis. The number of participants with TE substitutions in the spike protein reflects participants that had a TE change in the spike protein at any position including the sotrovimab epitope. AA substitutions compared to the reference strain are presented at Day 14.
Time Frame: At Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab 500 mg IV
Number analyzed (Participants) | 71
Participants
  AA substitutions >5% allelic frequency | 37
  AA substitutions >50% allelic frequency | 17

6. Primary Outcome: Number of Participants With Treatment Emergent Amino Acid Substitutions >5% and >50% Allelic Frequency in the Spike Protein at Day 28
Description: SARS-CoV-2 spike analysis was carried out by nucleotide sequencing of the SARS-CoV-2 spike protein by NGS analysis of participant nasal/oropharyngeal swab samples. The nucleotide sequences were translated, and the AA sequences aligned and compared to a reference sequence. Treatment emergent (TE) substitutions are defined as AA differences in a post-Baseline sample that were not present at Baseline at the defined threshold for minority and consensus analysis. The number of participants with TE substitutions in the spike protein reflects participants that had a TE change in the spike protein at any position including the sotrovimab epitope. AA substitutions compared to the reference strain are presented at Day 28.
Time Frame: At Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab 500 mg IV
Number analyzed (Participants) | 33
Participants
  AA substitutions >5% allelic frequency | 20
  AA substitutions >50% allelic frequency | 13

7. Secondary Outcome: Number of Participants With Variants of Concern (VOC) or Variants Under Investigation (VUI)
Description: SARS-CoV-2 VOC is defined by World health Organization(WHO) that meets definition of VUI and through a comparative assessment, has been demonstrated to be associated with 1 or more of following changes at degree of global public health(GPH) significance: increase in transmissibility or detrimental change in COVID-19 epidemiology, OR increase in virulence or change in clinical disease presentation, OR decrease in effectiveness of public health and social measures or available diagnostics, vaccines, therapeutics. SARS-CoV-2 VUI is defined by WHO as a variant:with genetic changes that are predicted or known to affect virus characteristics such as transmissibility, disease severity, immune, diagnostic or therapeutic escape and identified to cause significant community transmission or multiple COVID-19 clusters, in multiple countries with increasing relative prevalence alongside increasing number of cases over time, or other apparent epidemiological impacts to suggest emerging risk to GPH.
Time Frame: Up to Day 28
Population: The Safety Set included all participants who were enrolled and exposed to study intervention. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. Number of participants with any VOC/VUI based on WHO classification and Pango sub-lineage for the earliest possible VOC/VUI sample has been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab 500 mg IV
Number analyzed (Participants) | 208
Participants | 208

8. Secondary Outcome: Number of Participants With Undetectable Virus by Reverse Transcriptase Polymerase Chain Reaction (RT-PCR)
Description: The number of participants that had undetectable viral load in nasal/oropharyngeal swabs was determined by quantitative reverse transcription-polymerase chain reaction (qRT/PCR) at Day 7, Day 14, and Day 28. Participants with major protocol deviation (out of visit window/samples received late/return more samples than expected) at specific visits were excluded from analysis.
Time Frame: At Day 7, Day 14, and Day 28
Population: The Safety Set included all participants who were enrolled and exposed to study intervention, and represents the Overall Number of Participants Analyzed field (i.e., contributed data reported in the table). 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab 500 mg IV
Number analyzed (Participants) | 217
Participants
  Day 7: number analyzed (Participants) | 199
  Day 7 | 50
  Day 14: number analyzed (Participants) | 196
  Day 14 | 129
  Day 28: number analyzed (Participants) | 194
  Day 28 | 162

9. Secondary Outcome: Number of Participants With All Cause Hospital Stay
Description: Number of participants hospitalized due to any cause have been reported.
Time Frame: Up to Day 28
Population: The Safety Set included all participants who were enrolled and exposed to study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab 500 mg IV
Number analyzed (Participants) | 217
Participants | 7

10. Secondary Outcome: Number of Participants With COVID-19 Related Hospital Stay
Description: Number of participants hospitalized due to COVID-19 have been reported.
Time Frame: Up to Day 28
Population: The Safety Set included all participants who were enrolled and exposed to study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab 500 mg IV
Number analyzed (Participants) | 217
Participants | 0

11. Secondary Outcome: Number of Participants Requiring New or Increased Oxygen Support (Supplemental Oxygen [Not High Flow]), Non-invasive Ventilation or High-flow, Invasive Mechanical Ventilation or Extracorporeal Membrane Oxygenation (ECMO)
Description: Number of participants required new or increased oxygen support (supplemental oxygen [not high flow]), non-invasive ventilation or high-flow, invasive mechanical ventilation or ECMO have been reported.
Time Frame: Up to Day 28
Population: The Safety Set included all participants who were enrolled and exposed to study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab 500 mg IV
Number analyzed (Participants) | 217
Participants
  New or increased oxygen support (supplemental oxygen [not high flow]) | 1
  Non-invasive ventilation or high flow | 1
  Invasive mechanical ventilation | 0
  ECMO | 0

12. Secondary Outcome: Number of Participants With All Cause Intensive Care Unit (ICU) Hospital Stay
Description: Number of participants hospitalized in ICU due to any cause have been reported.
Time Frame: Up to Day 28
Population: The Safety Set included all participants who were enrolled and exposed to study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab 500 mg IV
Number analyzed (Participants) | 217
Participants | 0

13. Secondary Outcome: Number of Participants With COVID-19 Related ICU Hospital Stay
Description: Number of participants hospitalized in ICU due to COVID-19 have been reported.
Time Frame: Up to Day 28
Population: The Safety Set included all participants who were enrolled and exposed to study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab 500 mg IV
Number analyzed (Participants) | 217
Participants | 0

14. Secondary Outcome: Number of Participants Who Died Due to Any Cause Through Day 28
Description: Data for number of participants who died due to any cause through Day 28 have been reported.
Time Frame: Up to Day 28
Population: The Safety Set included all participants who were enrolled and exposed to study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab 500 mg IV
Number analyzed (Participants) | 217
Participants | 1

15. Secondary Outcome: Number of Participants Who Died Due to COVID-19 Through Day 28
Description: Data for number of participants who died due to COVID-19 have been reported.
Time Frame: Up to Day 28
Population: The Safety Set included all participants who were enrolled and exposed to study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab 500 mg IV
Number analyzed (Participants) | 217
Participants | 0

16. Secondary Outcome: Number of Participants With Treatment-emergent Amino Acid Substitutions in the Spike Protein for Any Substitutions at Allelic Frequency >5%
Description: SARS-CoV-2 spike analysis was carried out by nucleotide sequencing of the SARS-CoV-2 spike protein by NGS analysis of participant nasal/oropharyngeal swab samples for samples above the threshold for the sequencing assay. The nucleotide sequences were translated, and the AA sequences aligned and compared to a reference sequence. For samples with AA changes above the >5% threshold for allelic frequency determination, AA changes in SARS-CoV-2 spike protein compared to Baseline was reported. One participant may have more than one substitution under the same codon. Treatment Emergent Substitutions included participants where a Baseline and post-Baseline records exist. All type of AA mutations have been categorized.
Time Frame: At Day 7, Day 14 and Day 28
Population: The Safety Set included all participants who were enrolled and exposed to study intervention. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field, and represents participants who had Baseline and post-Baseline sequence available. 'Number Analyzed' signifies participants evaluable for the specified time points and codons at the >5% allelic frequency.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab 500 mg IV
Number analyzed (Participants) | 156
Participants
  Day 7, L5-L5F: number analyzed (Participants) | 142
  Day 7, L5-L5F | 1
  Day 7, L5-L5F Frameshift mutation: number analyzed (Participants) | 142
  Day 7, L5-L5F Frameshift mutation | 1
  Day 7, P39-P39L: number analyzed (Participants) | 141
  Day 7, P39-P39L | 1
  Day 7, G75-G75C: number analyzed (Participants) | 139
  Day 7, G75-G75C | 1
  Day 7, G75-G75V: number analyzed (Participants) | 139
  Day 7, G75-G75V | 1
  Day 7, T95-T95I: number analyzed (Participants) | 140
  Day 7, T95-T95I | 1
  Day 7, F106-F106 Deletion mutation: number analyzed (Participants) | 141
  Day 7, F106-F106 Deletion mutation | 1
  Day 7, Y144-Y144 Deletion mutation: number analyzed (Participants) | 114
  Day 7, Y144-Y144 Deletion mutation | 1
  Day 7, H146-H146Q Frameshift mutation: number analyzed (Participants) | 114
  Day 7, H146-H146Q Frameshift mutation | 1
  Day 7, V320-V320A: number analyzed (Participants) | 82
  Day 7, V320-V320A | 1
  Day 7, P330-P330S: number analyzed (Participants) | 85
  Day 7, P330-P330S | 2
  Day 7, P337-P337A: number analyzed (Participants) | 92
  Day 7, P337-P337A | 2
  Day 7, P337-P337H: number analyzed (Participants) | 92
  Day 7, P337-P337H | 2
  Day 7, P337-P337L: number analyzed (Participants) | 92
  Day 7, P337-P337L | 8
  Day 7, P337-P337R: number analyzed (Participants) | 92
  Day 7, P337-P337R | 2
  Day 7, P337-P337S: number analyzed (Participants) | 92
  Day 7, P337-P337S | 14
  Day 7, G339-G339R: number analyzed (Participants) | 91
  Day 7, G339-G339R | 1
  Day 7, G339-G339Y: number analyzed (Participants) | 91
  Day 7, G339-G339Y | 1
  Day 7, E340-E340A: number analyzed (Participants) | 91
  Day 7, E340-E340A | 3
  Day 7, E340-E340D: number analyzed (Participants) | 91
  Day 7, E340-E340D | 15
  Day 7, E340-E340G: number analyzed (Participants) | 91
  Day 7, E340-E340G | 5
  Day 7, E340-E340K: number analyzed (Participants) | 91
  Day 7, E340-E340K | 6
  Day 7, E340-E340Q: number analyzed (Participants) | 91
  Day 7, E340-E340Q | 14
  Day 7, E340-E340V: number analyzed (Participants) | 91
  Day 7, E340-E340V | 2
  Day 7, K356-K356M: number analyzed (Participants) | 90
  Day 7, K356-K356M | 1
  Day 7, K356-K356R: number analyzed (Participants) | 90
  Day 7, K356-K356R | 1
  Day 7, K356-K356T: number analyzed (Participants) | 90
  Day 7, K356-K356T | 6
  Day 7, S373-S373P: number analyzed (Participants) | 82
  Day 7, S373-S373P | 1
  Day 7, Q474-Q474 Deletion mutation: number analyzed (Participants) | 137
  Day 7, Q474-Q474 Deletion mutation | 1
  Day 7, Q493-Q493K: number analyzed (Participants) | 138
  Day 7, Q493-Q493K | 1
  Day 7, G496-G496V: number analyzed (Participants) | 137
  Day 7, G496-G496V | 1
  Day 7, V503-V503F: number analyzed (Participants) | 137
  Day 7, V503-V503F | 1
  Day 7, L517-L517F: number analyzed (Participants) | 136
  Day 7, L517-L517F | 1
  Day 7, L517-L517P: number analyzed (Participants) | 136
  Day 7, L517-L517P | 1
  Day 7, T523-T523I: number analyzed (Participants) | 136
  Day 7, T523-T523I | 1
  Day 7, F543-F543L: number analyzed (Participants) | 135
  Day 7, F543-F543L | 1
  Day 7, T547-T547K: number analyzed (Participants) | 135
  Day 7, T547-T547K | 1
  Day 7, K558-K558 Deletion mutation: number analyzed (Participants) | 149
  Day 7, K558-K558 Deletion mutation | 1
  Day 7, A570-A570T: number analyzed (Participants) | 149
  Day 7, A570-A570T | 1
  Day 7, T572-T572I: number analyzed (Participants) | 149
  Day 7, T572-T572I | 1
  Day 7, P579-P579L: number analyzed (Participants) | 149
  Day 7, P579-P579L | 1
  Day 7, L585-L585F: number analyzed (Participants) | 149
  Day 7, L585-L585F | 1
  Day 7, C590-C590Y: number analyzed (Participants) | 149
  Day 7, C590-C590Y | 1
  Day 7, F592-F592 Deletion mutation: number analyzed (Participants) | 148
  Day 7, F592-F592 Deletion mutation | 1
  Day 7, V622-V622I: number analyzed (Participants) | 145
  Day 7, V622-V622I | 1
  Day 7, H625- H625N: number analyzed (Participants) | 145
  Day 7, H625- H625N | 1
  Day 7, S640-S640F: number analyzed (Participants) | 145
  Day 7, S640-S640F | 1
  Day 7, Y660-Y660H: number analyzed (Participants) | 145
  Day 7, Y660-Y660H | 2
  Day 7, I666- I666 Deletion mutation: number analyzed (Participants) | 145
  Day 7, I666- I666 Deletion mutation | 1
  Day 7, G667-G667 Deletion mutation: number analyzed (Participants) | 145
  Day 7, G667-G667 Deletion mutation | 1
  Day 7, A668-A668 Deletion mutation: number analyzed (Participants) | 145
  Day 7, A668-A668 Deletion mutation | 1
  Day 7, G669-G669 Deletion mutation: number analyzed (Participants) | 145
  Day 7, G669-G669 Deletion mutation | 1
  Day 7, I670-I670 Deletion mutation: number analyzed (Participants) | 145
  Day 7, I670-I670 Deletion mutation | 1
  Day 7, C671-C671 Deletion mutation: number analyzed (Participants) | 145
  Day 7, C671-C671 Deletion mutation | 1
  Day 7, A672-A672 Deletion mutation: number analyzed (Participants) | 145
  Day 7, A672-A672 Deletion mutation | 1
  Day 7, S673-S673 Deletion mutation: number analyzed (Participants) | 145
  Day 7, S673-S673 Deletion mutation | 1
  Day 7, Y674-Y674 Deletion mutation: number analyzed (Participants) | 145
  Day 7, Y674-Y674 Deletion mutation | 1
  Day 7, Q675-Q675H: number analyzed (Participants) | 145
  Day 7, Q675-Q675H | 1
  Day 7, L752-L752F: number analyzed (Participants) | 78
  Day 7, L752-L752F | 1
  Day 7, N777-N777 Deletion mutation: number analyzed (Participants) | 136
  Day 7, N777-N777 Deletion mutation | 2
  Day 7, I794-I794T: number analyzed (Participants) | 136
  Day 7, I794-I794T | 1
  Day 7, L822-L822 Deletion mutation: number analyzed (Participants) | 135
  Day 7, L822-L822 Deletion mutation | 1
  Day 7, L822-L822F: number analyzed (Participants) | 135
  Day 7, L822-L822F | 1
  Day 7, F823-F823 Deletion mutation: number analyzed (Participants) | 135
  Day 7, F823-F823 Deletion mutation | 1
  Day 7, A845-A845V: number analyzed (Participants) | 135
  Day 7, A845-A845V | 1
  Day 7, A846-A846T: number analyzed (Participants) | 135
  Day 7, A846-A846T | 1
  Day 7, A846-A846V: number analyzed (Participants) | 135
  Day 7, A846-A846V | 1
  Day 7, I850-I850T: number analyzed (Participants) | 135
  Day 7, I850-I850T | 1
  Day 7, P862-P862S: number analyzed (Participants) | 135
  Day 7, P862-P862S | 1
  Day 7, Q913-Q913 Stop codon mutation: number analyzed (Participants) | 143
  Day 7, Q913-Q913 Stop codon mutation | 1
  Day 7, A930-A930 Deletion mutation: number analyzed (Participants) | 143
  Day 7, A930-A930 Deletion mutation | 1
  Day 7, Q954-Q954Y: number analyzed (Participants) | 143
  Day 7, Q954-Q954Y | 1
  Day 7, F970-F970L: number analyzed (Participants) | 145
  Day 7, F970-F970L | 1
  Day 7, S974-S974L: number analyzed (Participants) | 145
  Day 7, S974-S974L | 1
  Day 7, V987-V987F: number analyzed (Participants) | 145
  Day 7, V987-V987F | 1
  Day 7, A989-A989V: number analyzed (Participants) | 145
  Day 7, A989-A989V | 1
  Day 7, K1038-K1038E: number analyzed (Participants) | 137
  Day 7, K1038-K1038E | 1
  Day 7, C1043-C1043 Deletion mutation: number analyzed (Participants) | 137
  Day 7, C1043-C1043 Deletion mutation | 1
  Day 7, H1048-H1048Y: number analyzed (Participants) | 137
  Day 7, H1048-H1048Y | 1
  Day 7, L1049-L1049F: number analyzed (Participants) | 137
  Day 7, L1049-L1049F | 2
  Day 7, P1053-P1053S: number analyzed (Participants) | 137
  Day 7, P1053-P1053S | 1
  Day 7, H1058-H1058Y: number analyzed (Participants) | 137
  Day 7, H1058-H1058Y | 1
  Day 7, V1060-V1060I: number analyzed (Participants) | 137
  Day 7, V1060-V1060I | 1
  Day 7, F1103-F1103S: number analyzed (Participants) | 141
  Day 7, F1103-F1103S | 1
  Day 7, I1130-I1130L: number analyzed (Participants) | 136
  Day 7, I1130-I1130L | 1
  Day 7, D1146-D1146H: number analyzed (Participants) | 133
  Day 7, D1146-D1146H | 1
  Day 7, Q1208-Q1208 Stop codon mutation: number analyzed (Participants) | 141
  Day 7, Q1208-Q1208 Stop codon mutation | 1
  Day 7, Q1208-Q1208H: number analyzed (Participants) | 141
  Day 7, Q1208-Q1208H | 1
  Day 7, W1214-W1214C: number analyzed (Participants) | 141
  Day 7, W1214-W1214C | 1
  Day 7, F1220-F1220 Deletion mutation: number analyzed (Participants) | 141
  Day 7, F1220-F1220 Deletion mutation | 1
  Day 7, C1254-C1254 Stop codon mutation: number analyzed (Participants) | 139
  Day 7, C1254-C1254 Stop codon mutation | 20
  Day 7, E1258-E1258H: number analyzed (Participants) | 139
  Day 7, E1258-E1258H | 1
  Day 7, E1258-E1258Q: number analyzed (Participants) | 139
  Day 7, E1258-E1258Q | 1
  Day 7, P1263-P1263L: number analyzed (Participants) | 145
  Day 7, P1263-P1263L | 1
  Day 14, L5-L5F: number analyzed (Participants) | 55
  Day 14, L5-L5F | 1
  Day 14, L5-L5 Frameshift mutation: number analyzed (Participants) | 55
  Day 14, L5-L5 Frameshift mutation | 1
  Day 14, C15-C15F: number analyzed (Participants) | 57
  Day 14, C15-C15F | 1
  Day 14, Q23-Q23 Stop codon mutation: number analyzed (Participants) | 56
  Day 14, Q23-Q23 Stop codon mutation | 1
  Day 14, A67-A67V: number analyzed (Participants) | 53
  Day 14, A67-A67V | 1
  Day 14, F79-F79 Deletion mutation: number analyzed (Participants) | 54
  Day 14, F79-F79 Deletion mutation | 1
  Day 14, D88-D88G: number analyzed (Participants) | 54
  Day 14, D88-D88G | 1
  Day 14, E132-E132 Deletion mutation: number analyzed (Participants) | 44
  Day 14, E132-E132 Deletion mutation | 1
  Day 14, F133-F133 Deletion mutation: number analyzed (Participants) | 40
  Day 14, F133-F133 Deletion mutation | 1
  Day 14, D138-D138Y: number analyzed (Participants) | 39
  Day 14, D138-D138Y | 1
  Day 14, P139-P139 Deletion mutation: number analyzed (Participants) | 39
  Day 14, P139-P139 Deletion mutation | 2
  Day 14, F140-F140 Deletion mutation: number analyzed (Participants) | 39
  Day 14, F140-F140 Deletion mutation | 2
  Day 14, L141-L141 Deletion mutation: number analyzed (Participants) | 39
  Day 14, L141-L141 Deletion mutation | 2
  Day 14, G142-G142 Deletion mutation: number analyzed (Participants) | 39
  Day 14, G142-G142 Deletion mutation | 2
  Day 14, V143-V143 Deletion mutation: number analyzed (Participants) | 38
  Day 14, V143-V143 Deletion mutation | 2
  Day 14, Y144-Y144 Deletion mutation: number analyzed (Participants) | 39
  Day 14, Y144-Y144 Deletion mutation | 3
  Day 14, Y145-Y145 Deletion mutation: number analyzed (Participants) | 38
  Day 14, Y145-Y145 Deletion mutation | 1
  Day 14, H146-H146 Deletion mutation: number analyzed (Participants) | 38
  Day 14, H146-H146 Deletion mutation | 1
  Day 14, H146-H146Y: number analyzed (Participants) | 38
  Day 14, H146-H146Y | 1
  Day 14, W152-W152L: number analyzed (Participants) | 37
  Day 14, W152-W152L | 1
  Day 14, M153-M153I: number analyzed (Participants) | 37
  Day 14, M153-M153I | 1
  Day 14, A243-A243 Deletion mutation: number analyzed (Participants) | 3
  Day 14, A243-A243 Deletion mutation | 1
  Day 14, L244-L244 Deletion mutation: number analyzed (Participants) | 3
  Day 14, L244-L244 Deletion mutation | 1
  Day 14, P337-P337H: number analyzed (Participants) | 26
  Day 14, P337-P337H | 1
  Day 14, P337-P337L: number analyzed (Participants) | 26
  Day 14, P337-P337L | 4
  Day 14, P337-P337R: number analyzed (Participants) | 26
  Day 14, P337-P337R | 1
  Day 14, P337-P337S: number analyzed (Participants) | 26
  Day 14, P337-P337S | 6
  Day 14, E340-E340D: number analyzed (Participants) | 26
  Day 14, E340-E340D | 5
  Day 14, E340-E340G: number analyzed (Participants) | 26
  Day 14, E340-E340G | 4
  Day 14, E340-E340K: number analyzed (Participants) | 26
  Day 14, E340-E340K | 5
  Day 14, E340-E340Q: number analyzed (Participants) | 26
  Day 14, E340-E340Q | 7
  Day 14, E340-E340V: number analyzed (Participants) | 26
  Day 14, E340-E340V | 2
  Day 14, R346-R346T: number analyzed (Participants) | 26
  Day 14, R346-R346T | 1
  Day 14, K356-K356T: number analyzed (Participants) | 26
  Day 14, K356-K356T | 1
  Day 14, T376-T376 Deletion mutation: number analyzed (Participants) | 26
  Day 14, T376-T376 Deletion mutation | 1
  Day 14, F377-F377 Deletion mutation: number analyzed (Participants) | 26
  Day 14, F377-F377 Deletion mutation | 1
  Day 14, K444-K444S: number analyzed (Participants) | 20
  Day 14, K444-K444S | 1
  Day 14, V503-V503A: number analyzed (Participants) | 48
  Day 14, V503-V503A | 1
  Day 14, Y505-Y505N: number analyzed (Participants) | 48
  Day 14, Y505-Y505N | 1
  Day 14, R509-R509T: number analyzed (Participants) | 48
  Day 14, R509-R509T | 1
  Day 14, K528-K528E: number analyzed (Participants) | 46
  Day 14, K528-K528E | 1
  Day 14, T547-T547K: number analyzed (Participants) | 46
  Day 14, T547-T547K | 1
  Day 14, A570-A570T: number analyzed (Participants) | 62
  Day 14, A570-A570T | 1
  Day 14, T572-T572I: number analyzed (Participants) | 62
  Day 14, T572-T572I | 1
  Day 14, D574-D574N: number analyzed (Participants) | 62
  Day 14, D574-D574N | 1
  Day 14, L611-L611P: number analyzed (Participants) | 56
  Day 14, L611-L611P | 1
  Day 14, G639-G639V: number analyzed (Participants) | 56
  Day 14, G639-G639V | 1
  Day 14, G669-G669 Deletion mutation: number analyzed (Participants) | 56
  Day 14, G669-G669 Deletion mutation | 1
  Day 14, I670-I670N: number analyzed (Participants) | 56
  Day 14, I670-I670N | 1
  Day 14, C671-C671 Deletion mutation: number analyzed (Participants) | 56
  Day 14, C671-C671 Deletion mutation | 1
  Day 14, A672-A672 Deletion mutation: number analyzed (Participants) | 56
  Day 14, A672-A672 Deletion mutation | 1
  Day 14, S673-S673 Deletion mutation: number analyzed (Participants) | 56
  Day 14, S673-S673 Deletion mutation | 1
  Day 14, Y674-Y674 Deletion mutation: number analyzed (Participants) | 56
  Day 14, Y674-Y674 Deletion mutation | 1
  Day 14, Q675-Q675H: number analyzed (Participants) | 56
  Day 14, Q675-Q675H | 1
  Day 14, A694-A694S: number analyzed (Participants) | 23
  Day 14, A694-A694S | 1
  Day 14, T859-T859 Deletion mutation: number analyzed (Participants) | 48
  Day 14, T859-T859 Deletion mutation | 1
  Day 14, V860-V860 Deletion mutation: number analyzed (Participants) | 48
  Day 14, V860-V860 Deletion mutation | 1
  Day 14, A879-A879V: number analyzed (Participants) | 58
  Day 14, A879-A879V | 1
  Day 14, A893-A893S: number analyzed (Participants) | 59
  Day 14, A893-A893S | 1
  Day 14, K921-K921 Deletion mutation: number analyzed (Participants) | 55
  Day 14, K921-K921 Deletion mutation | 1
  Day 14, V951-V951L: number analyzed (Participants) | 53
  Day 14, V951-V951L | 1
  Day 14, A956-A956E: number analyzed (Participants) | 53
  Day 14, A956-A956E | 1
  Day 14, V987-V987F: number analyzed (Participants) | 59
  Day 14, V987-V987F | 1
  Day 14, R1019-R1019I Frameshift mutation: number analyzed (Participants) | 52
  Day 14, R1019-R1019I Frameshift mutation | 1
  Day 14, Y1067-Y1067H: number analyzed (Participants) | 57
  Day 14, Y1067-Y1067H | 1
  Day 14, F1089-F1089S: number analyzed (Participants) | 55
  Day 14, F1089-F1089S | 1
  Day 14, F1095-F1095L: number analyzed (Participants) | 47
  Day 14, F1095-F1095L | 1
  Day 14, E1150-E1150G: number analyzed (Participants) | 44
  Day 14, E1150-E1150G | 1
  Day 14, M1229-M1229I: number analyzed (Participants) | 50
  Day 14, M1229-M1229I | 1
  Day 14, L1244-L1244 Deletion mutation: number analyzed (Participants) | 50
  Day 14, L1244-L1244 Deletion mutation | 1
  Day 14, K1245-K1245 Stop codon mutation: number analyzed (Participants) | 50
  Day 14, K1245-K1245 Stop codon mutation | 1
  Day 14, C1254-C1254 Stop codon mutation: number analyzed (Participants) | 50
  Day 14, C1254-C1254 Stop codon mutation | 7
  Day 28, F32-F32 Deletion mutation: number analyzed (Participants) | 24
  Day 28, F32-F32 Deletion mutation | 1
  Day 28, R78-R78S: number analyzed (Participants) | 22
  Day 28, R78-R78S | 1
  Day 28, F133-F133S: number analyzed (Participants) | 18
  Day 28, F133-F133S | 1
  Day 28, D138-D138Y: number analyzed (Participants) | 18
  Day 28, D138-D138Y | 1
  Day 28, P139-P139 Deletion mutation: number analyzed (Participants) | 18
  Day 28, P139-P139 Deletion mutation | 1
  Day 28, F140-F140 Deletion mutation: number analyzed (Participants) | 18
  Day 28, F140-F140 Deletion mutation | 1
  Day 28, L141-L141 Deletion mutation: number analyzed (Participants) | 18
  Day 28, L141-L141 Deletion mutation | 1
  Day 28, G142-G142 Deletion mutation: number analyzed (Participants) | 18
  Day 28, G142-G142 Deletion mutation | 1
  Day 28, V143-V143 Deletion mutation: number analyzed (Participants) | 18
  Day 28, V143-V143 Deletion mutation | 1
  Day 28, Y144-Y144 Deletion mutation: number analyzed (Participants) | 18
  Day 28, Y144-Y144 Deletion mutation | 5
  Day 28, Y145-Y145 Deletion mutation: number analyzed (Participants) | 18
  Day 28, Y145-Y145 Deletion mutation | 1
  Day 28, H146-H146 Deletion mutation: number analyzed (Participants) | 18
  Day 28, H146-H146 Deletion mutation | 1
  Day 28, N148-N148 Deletion mutation: number analyzed (Participants) | 18
  Day 28, N148-N148 Deletion mutation | 1
  Day 28, I210-I210N: number analyzed (Participants) | 18
  Day 28, I210-I210N | 1
  Day 28, N211-N211 Deletion mutation: number analyzed (Participants) | 18
  Day 28, N211-N211 Deletion mutation | 1
  Day 28, P330-P330S: number analyzed (Participants) | 12
  Day 28, P330-P330S | 1
  Day 28, P337-P337H: number analyzed (Participants) | 13
  Day 28, P337-P337H | 1
  Day 28, P337-P337S: number analyzed (Participants) | 13
  Day 28, P337-P337S | 2
  Day 28, E340-E340A: number analyzed (Participants) | 13
  Day 28, E340-E340A | 1
  Day 28, E340-E340D: number analyzed (Participants) | 13
  Day 28, E340-E340D | 1
  Day 28, E340-E340G: number analyzed (Participants) | 13
  Day 28, E340-E340G | 2
  Day 28, E340-E340K: number analyzed (Participants) | 13
  Day 28, E340-E340K | 1
  Day 28, E340-E340Q: number analyzed (Participants) | 13
  Day 28, E340-E340Q | 4
  Day 28, E340-E340V: number analyzed (Participants) | 13
  Day 28, E340-E340V | 2
  Day 28, K356-K356R: number analyzed (Participants) | 12
  Day 28, K356-K356R | 1
  Day 28, K356-K356T: number analyzed (Participants) | 12
  Day 28, K356-K356T | 1
  Day 28, T376-T376 Deletion mutation: number analyzed (Participants) | 10
  Day 28, T376-T376 Deletion mutation | 1
  Day 28, F377-F377 Deletion mutation: number analyzed (Participants) | 11
  Day 28, F377-F377 Deletion mutation | 1
  Day 28, D420-D420N: number analyzed (Participants) | 7
  Day 28, D420-D420N | 1
  Day 28, G446-G446D: number analyzed (Participants) | 5
  Day 28, G446-G446D | 1
  Day 28, G446-G446R: number analyzed (Participants) | 5
  Day 28, G446-G446R | 1
  Day 28, G476-G476R: number analyzed (Participants) | 22
  Day 28, G476-G476R | 1
  Day 28, N481-N481K: number analyzed (Participants) | 22
  Day 28, N481-N481K | 1
  Day 28, Y489-Y489H: number analyzed (Participants) | 22
  Day 28, Y489-Y489H | 1
  Day 28, G496-G496V: number analyzed (Participants) | 22
  Day 28, G496-G496V | 1
  Day 28, Y505-Y505N: number analyzed (Participants) | 22
  Day 28, Y505-Y505N | 1
  Day 28, L513-L513F: number analyzed (Participants) | 22
  Day 28, L513-L513F | 1
  Day 28, L517-L517F: number analyzed (Participants) | 22
  Day 28, L517-L517F | 1
  Day 28, T547-T547K: number analyzed (Participants) | 22
  Day 28, T547-T547K | 1
  Day 28, T572-T572I: number analyzed (Participants) | 25
  Day 28, T572-T572I | 1
  Day 28, S591-S591F: number analyzed (Participants) | 25
  Day 28, S591-S591F | 1
  Day 28, G593-G593V: number analyzed (Participants) | 25
  Day 28, G593-G593V | 1
  Day 28, P631-P631S: number analyzed (Participants) | 24
  Day 28, P631-P631S | 1
  Day 28, Q644-Q644 Frameshift mutation: number analyzed (Participants) | 24
  Day 28, Q644-Q644 Frameshift mutation | 1
  Day 28, A647-A647S: number analyzed (Participants) | 24
  Day 28, A647-A647S | 1
  Day 28, Q675-Q675H: number analyzed (Participants) | 24
  Day 28, Q675-Q675H | 1
  Day 28, T676-T676I: number analyzed (Participants) | 24
  Day 28, T676-T676I | 1
  Day 28, K795-K795 Deletion mutation: number analyzed (Participants) | 23
  Day 28, K795-K795 Deletion mutation | 1
  Day 28, Q872-Q872 Stop codon mutation: number analyzed (Participants) | 21
  Day 28, Q872-Q872 Stop codon mutation | 1
  Day 28, T883-T883I: number analyzed (Participants) | 25
  Day 28, T883-T883I | 1
  Day 28, A899-A899C Frameshift mutation: number analyzed (Participants) | 24
  Day 28, A899-A899C Frameshift mutation | 1
  Day 28, D979-D979V: number analyzed (Participants) | 25
  Day 28, D979-D979V | 1
  Day 28, V987-V987F: number analyzed (Participants) | 25
  Day 28, V987-V987F | 1
  Day 28, Q1002-Q1002 Stop codon mutation: number analyzed (Participants) | 24
  Day 28, Q1002-Q1002 Stop codon mutation | 1
  Day 28, A1020-A1020V: number analyzed (Participants) | 24
  Day 28, A1020-A1020V | 1
  Day 28, H1048-H1048Y: number analyzed (Participants) | 24
  Day 28, H1048-H1048Y | 1
  Day 28, F1103-F1103V: number analyzed (Participants) | 23
  Day 28, F1103-F1103V | 1
  Day 28, T1117-T1117I: number analyzed (Participants) | 23
  Day 28, T1117-T1117I | 1
  Day 28, S1123-S1123P: number analyzed (Participants) | 23
  Day 28, S1123-S1123P | 1
  Day 28, I1227-I1227 Deletion mutation: number analyzed (Participants) | 23
  Day 28, I1227-I1227 Deletion mutation | 1
  Day 28, C1254-C1254 Stop codon mutation: number analyzed (Participants) | 22
  Day 28, C1254-C1254 Stop codon mutation | 5

17. Secondary Outcome: Number of Participants With Treatment-emergent Amino Acid Substitutions in the Spike Protein for Any Substitutions at Allelic Frequency >50%
Description: SARS-CoV-2 spike analysis was carried out by nucleotide sequencing of the SARS-CoV-2 spike protein by NGS analysis of participant nasal/oropharyngeal swab samples for samples with viral load above the threshold of the sequencing assay. The nucleotide sequences were translated, and the AA sequences aligned and compared to a reference sequence. For samples with AA changes above the threshold for consensus sequence generation that were not present in the Baseline sequence, AA changes in the SARS-CoV-2 spike protein consensus sequence (>50%) from Baseline was reported. One participant may have more than one substitution under the same codon. Treatment Emergent Substitutions included participants where a Baseline and post-Baseline records exist. All type of AA mutations have been categorized.
Time Frame: At Day 7, Day 14 and Day 28
Population: The Safety Set included all participants who were enrolled and exposed to study intervention. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field, and represents participants who had Baseline and post-Baseline sequence available. 'Number Analyzed' signifies participants evaluable for the specified time points and codons at the >50% allelic frequency.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotrovimab 500 mg IV
Number analyzed (Participants) | 156
Participants
  Day 7, G75-G75V: number analyzed (Participants) | 139
  Day 7, G75-G75V | 1
  Day 7, P337-P337L: number analyzed (Participants) | 92
  Day 7, P337-P337L | 1
  Day 7, P337-P337S: number analyzed (Participants) | 92
  Day 7, P337-P337S | 3
  Day 7, E340-E340A: number analyzed (Participants) | 91
  Day 7, E340-E340A | 1
  Day 7, E340-E340D: number analyzed (Participants) | 91
  Day 7, E340-E340D | 2
  Day 7, E340-E340G: number analyzed (Participants) | 91
  Day 7, E340-E340G | 1
  Day 7, E340-E340K: number analyzed (Participants) | 91
  Day 7, E340-E340K | 1
  Day 7, E340-E340Q: number analyzed (Participants) | 91
  Day 7, E340-E340Q | 3
  Day 7, S373-S373P: number analyzed (Participants) | 82
  Day 7, S373-S373P | 1
  Day 7, Q675-Q675H: number analyzed (Participants) | 145
  Day 7, Q675-Q675H | 1
  Day 7, L752-L752F: number analyzed (Participants) | 78
  Day 7, L752-L752F | 1
  Day 7, A845-A845V: number analyzed (Participants) | 135
  Day 7, A845-A845V | 1
  Day 7, A846-A846T: number analyzed (Participants) | 135
  Day 7, A846-A846T | 1
  Day 7, Q913-Q913 Stop codon mutation: number analyzed (Participants) | 143
  Day 7, Q913-Q913 Stop codon mutation | 1
  Day 7, P1053-P1053S: number analyzed (Participants) | 137
  Day 7, P1053-P1053S | 1
  Day 14, L5-L5F: number analyzed (Participants) | 55
  Day 14, L5-L5F | 1
  Day 14, Y144-Y144 Deletion mutation: number analyzed (Participants) | 39
  Day 14, Y144-Y144 Deletion mutation | 1
  Day 14, P337-P337L: number analyzed (Participants) | 26
  Day 14, P337-P337L | 1
  Day 14, P337-P337S: number analyzed (Participants) | 26
  Day 14, P337-P337S | 1
  Day 14, E340-E340D: number analyzed (Participants) | 26
  Day 14, E340-E340D | 3
  Day 14, E340-E340K: number analyzed (Participants) | 26
  Day 14, E340-E340K | 1
  Day 14, E340-E340Q: number analyzed (Participants) | 26
  Day 14, E340-E340Q | 3
  Day 14, E340-E340V: number analyzed (Participants) | 26
  Day 14, E340-E340V | 1
  Day 14, K356-K356T: number analyzed (Participants) | 26
  Day 14, K356-K356T | 1
  Day 14, V503-V503A: number analyzed (Participants) | 48
  Day 14, V503-V503A | 1
  Day 14, Y505-Y505N: number analyzed (Participants) | 48
  Day 14, Y505-Y505N | 1
  Day 14, A570-A570T: number analyzed (Participants) | 62
  Day 14, A570-A570T | 1
  Day 14, T572-T572I: number analyzed (Participants) | 62
  Day 14, T572-T572I | 1
  Day 14, D574-D574N: number analyzed (Participants) | 62
  Day 14, D574-D574N | 1
  Day 14, I670- I670N: number analyzed (Participants) | 56
  Day 14, I670- I670N | 1
  Day 14, C671-C671 Deletion mutation: number analyzed (Participants) | 56
  Day 14, C671-C671 Deletion mutation | 1
  Day 14, A672-A672 Deletion mutation: number analyzed (Participants) | 56
  Day 14, A672-A672 Deletion mutation | 1
  Day 14, S673-S673 Deletion mutation: number analyzed (Participants) | 56
  Day 14, S673-S673 Deletion mutation | 1
  Day 14, Y674-Y674 Deletion mutation: number analyzed (Participants) | 56
  Day 14, Y674-Y674 Deletion mutation | 1
  Day 14, A956-A956E: number analyzed (Participants) | 53
  Day 14, A956-A956E | 1
  Day 14, L1244-L1244 Deletion mutation: number analyzed (Participants) | 50
  Day 14, L1244-L1244 Deletion mutation | 1
  Day 28, Y144-Y144 Deletion mutation: number analyzed (Participants) | 18
  Day 28, Y144-Y144 Deletion mutation | 3
  Day 28, I210-I210N: number analyzed (Participants) | 18
  Day 28, I210-I210N | 1
  Day 28, N211-N211 Deletion mutation: number analyzed (Participants) | 18
  Day 28, N211-N211 Deletion mutation | 1
  Day 28, P337-P337S: number analyzed (Participants) | 13
  Day 28, P337-P337S | 2
  Day 28, E340-E340A: number analyzed (Participants) | 13
  Day 28, E340-E340A | 1
  Day 28, E340-E340D: number analyzed (Participants) | 13
  Day 28, E340-E340D | 1
  Day 28, E340-E340G: number analyzed (Participants) | 13
  Day 28, E340-E340G | 1
  Day 28, E340-E340K: number analyzed (Participants) | 13
  Day 28, E340-E340K | 1
  Day 28, E340-E340Q: number analyzed (Participants) | 13
  Day 28, E340-E340Q | 3
  Day 28, E340-E340V: number analyzed (Participants) | 13
  Day 28, E340-E340V | 1
  Day 28, K356-K356R: number analyzed (Participants) | 12
  Day 28, K356-K356R | 1
  Day 28, D420-D420N: number analyzed (Participants) | 7
  Day 28, D420-D420N | 1
  Day 28, G446-G446D: number analyzed (Participants) | 5
  Day 28, G446-G446D | 1
  Day 28, N481-N481K: number analyzed (Participants) | 22
  Day 28, N481-N481K | 1
  Day 28, T572-T572I: number analyzed (Participants) | 25
  Day 28, T572-T572I | 1
  Day 28, P631-P631S: number analyzed (Participants) | 24
  Day 28, P631-P631S | 1
  Day 28, A647-A647S: number analyzed (Participants) | 24
  Day 28, A647-A647S | 1
  Day 28, T676-T676I: number analyzed (Participants) | 24
  Day 28, T676-T676I | 1
  Day 28, Q1002-Q1002 Stop codon mutation: number analyzed (Participants) | 24
  Day 28, Q1002-Q1002 Stop codon mutation | 1

ADVERSE EVENTS:
Time Frame: Up to Day 28
Description: All-cause mortality, Treatment-emergent serious adverse events (TESAEs) and Treatment-emergent non-SAEs were reported for the Safety Set (Safety Set included all participants who were enrolled and exposed to study intervention).
Arm/Group | Sotrovimab 500 mg IV
All-Cause Mortality (participants affected / at risk) | 1/217
Serious Adverse Events (participants affected / at risk) | 0/217
Other Adverse Events (participants affected / at risk) | 6/217
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sotrovimab 500 mg IV (N=217)
Diarrhoea (Gastrointestinal disorders) | 1
Blood creatinine increased (Investigations) | 1
Neutrophil count increased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Ageusia (Nervous system disorders) | 1
Anosmia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT05305651/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT05305651/SAP_001.pdf